CLINICAL TRIAL: NCT06463626
Title: REal-world Patterns of Treatment With CDKi 4/6 for AdVanced BrEast CAncer in PortugaL - REVEAL Study
Brief Title: Real-life Treatment Patterns With Cyclin-dependent Kinase Inhibitors in Advanced Breast Cancer in Portugal - REVEAL Study
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CLEE011APT01
Record Dates: First submitted 2024-06-10; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Hormone-receptor-positive Breast Cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- CDKi cohort: Adult women with HR-positive and HER-2-negative advanced breast cancer who started first- or second-line treatment with CDKi 4/6 (ribociclib or palbociclib).

SUMMARY:
This was a non-interventional (observational), retrospective, cohort study of women with hormone receptor (HR)-positive and human epidermal growth factor receptor-type 2 (HER2)-negative advanced breast cancer who started treatment with cyclin-dependent kinase inhibitors (CDKi) 4/6 (ribociclib or palbociclib) in Portugal. This was a study of medication use patterns, based on information from the hospital pharmacies of the participating centers.

Patients who started a CDKi 4/6 (ribociclib or palbociclib) between 1 March 2019 and 31 December 2019 were included and followed through 24 months. A follow-up occurred 6 months after the start of CDKi 4/6 (ribociclib or palbociclib) to quantify the occurrence of dose changes.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Aged 18 years or older at the time of starting therapy with CDKi 4/6.
* Breast cancer diagnosis.
* At least one record of ribociclib or palbociclib donation during the identification period.
* Registration of the first supply of ribociclib or palbociclib between 1 March 2019 and 31 December 2019.

Exclusion Criteria:

* Patients with missing information regarding their date of birth and the date or quantity of the drug dispensed in any assignment were excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Mean Age | Baseline, defined as start of treatment with CDKi
Number of Pre-menopause Patients by CDKi 4/6 | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Post-menopause Patients by CDKi 4/6 | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Patients Starting First-Line Therapy with CDKi 4/6 | Baseline, defined as start of treatment with CDKi
  Line of therapy: first-line therapy for advanced breast cancer was defined as no previous hormonal treatment in the 12 months prior to starting treatment with CDKi, including patients with concomitant treatment with fulvestrant. Second-line therapy was defined as previous hormonal treatment in the 12 months prior to starting treatment with CDKi.
Number of Patients Starting Second-Line Therapy with CDKi 4/6 | Baseline, defined as start of treatment with CDKi
  Line of therapy: first-line therapy for advanced breast cancer was defined as no previous hormonal treatment in the 12 months prior to starting treatment with CDKi, including patients with concomitant treatment with fulvestrant. Second-line therapy was defined as previous hormonal treatment in the 12 months prior to starting treatment with CDKi.
Initial Dose of CDKi 4/6 | Baseline, defined as start of treatment with CDKi
Number of Patients Administered Initial Dose of CDKi 4/6 Once per Day | Baseline, defined as start of treatment with CDKi
Number of Patients Without Concomitant Therapy | Baseline, defined as start of treatment with CDKi
Number of Palbociclib-treated Patients by Type of Concomitant Therapy | Baseline, defined as start of treatment with CDKi
Number of Ribociclib-treated Patients by Type of Concomitant Therapy | Baseline, defined as start of treatment with CDKi
Number of Palbociclib-treated Patients by Type of Aromatase Inhibitor | Baseline, defined as start of treatment with CDKi
Number of Ribociclib-treated Patients by Type of Aromatase Inhibitor | Baseline, defined as start of treatment with CDKi
Number of Pre-menopause Patients Without Concomitant Therapy | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Post-menopause Patients Without Concomitant Therapy | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Pre-menopause, Palbociclib-treated Patients by Type of Concomitant Therapy | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Pre-menopause, Ribociclib-treated Patients by Type of Concomitant Therapy | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Post-menopause, Palbociclib-treated Patients by Type of Concomitant Therapy | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Post-menopause, Ribociclib-treated Patients by Type of Concomitant Therapy | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Pre-menopause, Palbociclib-treated Patients by Type of Aromatase Inhibitor | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Pre-menopause, Ribociclib-treated Patients by Type of Aromatase Inhibitor | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Post-menopause, Palbociclib-treated Patients by Type of Aromatase Inhibitor | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.
Number of Post-menopause, Ribociclib-treated Patients by Type of Aromatase Inhibitor | Baseline, defined as start of treatment with CDKi
  Menopausal status: if the patient had taken goserelin in the six months before or after starting CDKi, she was considered to be pre-menopausal. In patients without an associated goserelin withdrawal, age was taken into account, and patients aged 50 or over were considered post-menopausal.

SECONDARY OUTCOMES:
Number of Patients with at Least One Dose Change | Up to 6 months post-initiation of CDKi treatment
Average Number of Dose Changes Per Patient | Up to 6 months post-initiation of CDKi treatment
Number of Palbociclib-treated Patients by Number of Dose Changes | Up to 6 months post-initiation of CDKi treatment
Number of Ribociclib-treated Patients by Number of Dose Changes | Up to 6 months post-initiation of CDKi treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States